CLINICAL TRIAL: NCT00398684
Title: Nevirapine Plus Zidovudine to Prevent Perinatal HIV in Thailand
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Harvard School of Public Health (HSPH) (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHPT-2; R01-HD39615; ANRS 1208
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections; Pregnancy
Keywords: Thailand; Developing countries; prophylaxis; mother to child transmission; HIV-1; HIV-1 infection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

ARMS (3):
- 1 (Experimental): One dose maternal NVP treatment at onset of labor, and one dose of infant NVP treatment 48-72 hours after birth (NVP-NVP)
  Interventions: Drug: Single dose nevirapine to the mother and to the child
- 2 (Experimental): One dose maternal NVP treatment at onset of labor, and one dose of infant placebo 48-72 hours after birth. (NVP-Placebo)
  Interventions: Drug: Single dose nevirapine to the mother and placebo to the child
- 3 (Placebo Comparator): One dose maternal placebo at onset of labor, and one dose of infant placebo 48-72 hours after birth. This was the reference study arm. (Placebo-Placebo)
  Interventions: Drug: Single dose placebo to the mother and to the child

INTERVENTIONS:
Drug: Single dose nevirapine to the mother and to the child — One maternal 200 mg NVP dose at the onset of labor, and one dose of infant NVP (0.6 ml/6mg) between 48-72 hours after birth. [Infants less than 2,500g received only 0.2mL/kg]
  Arms: 1
Drug: Single dose nevirapine to the mother and placebo to the child — One maternal 200 mg NVP dose at the onset of labor, and one dose of infant placebo (0.6 ml) between 48-72 hours after birth. [Infants less than 2,500g received only 0.2mL/kg]
  Arms: 2
Drug: Single dose placebo to the mother and to the child — One maternal placebo dose at the onset of labor, and one dose of infant placebo (0.6 ml) between 48-72 hours after birth. [Infants less than 2,500g received only 0.2mL/kg]
  Arms: 3

SUMMARY:
The purpose of this study was to assess the efficacy of a single dose of the drug nevirapine (NVP) given to pregnant women at onset of labor and to their infant 48-72 hours after birth in addition to standard oral zidovudine (ZDV or AZT) prophylaxis for the prevention of mother-to-child transmission of HIV-1.

DETAILED DESCRIPTION:
Multicenter, randomized, three arms, double-blind, controlled study. Study population was HIV-infected pregnant women who were on ZDV prophylaxis for more than two weeks and gave informed consent. If eligible, women completed a baseline check-up. Women meeting selection criteria were randomly assigned to receive one of three study regimens, in addition to ZDV prophylaxis:

1. One dose maternal NVP treatment at onset of labor, and one dose of infant NVP treatment 48-72 hours after birth
2. One dose maternal NVP treatment at onset of labor, and one dose of infant placebo 48-72 hours after birth
3. One dose maternal placebo at onset of labor, and one dose of infant placebo 48-72 hours after birth. This was the reference study arm.

Follow-up of women and infants was carried out on an outpatient basis except for delivery and the first three days after delivery.

AMENDMENT

After the first interim analysis, enrollment in Placebo-Placebo arm was terminated on May 2, 2002, according to the recommendation of the Data and Safety Monitoring Board. The target sample size was increased to 660, instead of 510, in each of the two remaining arms (N-N and N-P) to ensure enough power to test for non-inferiority between these arms with a limit of 2.5%.

ELIGIBILITY:
Pre-Entry Criteria

Women were eligible for the study if they:

* have evidence of HIV infection (documented by two HIV antibody tests on two different dates);
* were to be provided ZDV Prophylaxis (starting at 28 weeks or as soon as possible thereafter);
* intended to carry the pregnancy to term;
* intended to deliver at and bring their infant to a study site for at least 12 months after delivery; and
* could provide informed consent.

Inclusion criteria

Women are eligible for the study if they:

* met all pre-entry criteria;
* agreed not to breastfeed;
* consented to participate and to be followed for the duration of the study;
* presented the following laboratory values within 14 days prior to randomization:
* hemoglobin > 8.0 mg/dl
* absolute neutrophil count > 1000 cells/mm3
* platelets > 100,000 cells/mm3
* serum creatinine < 1.5 mg/dl (women with a serum creatinine > 1.5 mg/dl must have a measured eight-hour urine creatinine clearance > 70 ml/min)
* SGPT less than 10 times the upper limit of normal NOTE: Women with a Grade 2 or Grade 3 SGPT value (between 2.6 and 10 times the upper limit of normal) were allowed on study; they were monitored monthly until delivery. If at any point their SGPT value rose to a Grade 4 (more than 10 times the upper limit of normal), they should not be dosed with the Study Drug.

Exclusion Criteria:

* evidence of pre-existing fetal anomalies incompatible with life;
* known hypersensitivity to any benzodiazepine or to NVP;
* receipt of antiretroviral agent other than ZDV;
* receipt of non-allowed concomitant treatment;
* uncontrolled hypertension;
* concurrent participation in another clinical trial;
* women with a CD4 count <200/µL or history of oral candidiasis if they were not receiving PCP prophylaxis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1792
Dates: Start 2001-01; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Definitive HIV infection in infants as assessed by positive HIV DNA PCR on two peripheral blood samples

SECONDARY OUTCOMES:
Tolerance of nevirapine, in particular rashes.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lallemant, MD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (1):
- Phpt - Ird 174, Chiang Mai, Chiang Mai, Thailand

REFERENCES:
- [Background] Cressey TR, Jourdain G, Lallemant MJ, Kunkeaw S, Jackson JB, Musoke P, Capparelli E, Mirochnick M. Persistence of nevirapine exposure during the postpartum period after intrapartum single-dose nevirapine in addition to zidovudine prophylaxis for the prevention of mother-to-child transmission of HIV-1. J Acquir Immune Defic Syndr. 2005 Mar 1;38(3):283-8. PMID 15735445
- [Background] Jourdain G, Ngo-Giang-Huong N, Le Coeur S, Bowonwatanuwong C, Kantipong P, Leechanachai P, Ariyadej S, Leenasirimakul P, Hammer S, Lallemant M; Perinatal HIV Prevention Trial Group. Intrapartum exposure to nevirapine and subsequent maternal responses to nevirapine-based antiretroviral therapy. N Engl J Med. 2004 Jul 15;351(3):229-40. doi: 10.1056/NEJMoa041305. Epub 2004 Jul 9. PMID 15247339
- [Result] Lallemant M, Jourdain G, Le Coeur S, Mary JY, Ngo-Giang-Huong N, Koetsawang S, Kanshana S, McIntosh K, Thaineua V; Perinatal HIV Prevention Trial (Thailand) Investigators. Single-dose perinatal nevirapine plus standard zidovudine to prevent mother-to-child transmission of HIV-1 in Thailand. N Engl J Med. 2004 Jul 15;351(3):217-28. doi: 10.1056/NEJMoa033500. Epub 2004 Jul 9. PMID 15247338
- [Derived] Sripan P, Le Coeur S, Amzal B, Ingsrisawang L, Traisathit P, Ngo-Giang-Huong N, McIntosh K, Cressey TR, Sangsawang S, Rawangban B, Kanjanavikai P, Treluyer JM, Jourdain G, Lallemant M, Urien S. Modeling of In-Utero and Intra-Partum Transmissions to Evaluate the Efficacy of Interventions for the Prevention of Perinatal HIV. PLoS One. 2015 May 19;10(5):e0126647. doi: 10.1371/journal.pone.0126647. eCollection 2015. Erratum In: PLoS One. 2015 Jun 26;10(6):e0130917. doi: 10.1371/journal.pone.0130917. PLoS One. 2015 Aug 28;10(8):e0137368. doi: 10.1371/journal.pone.0137368. PMID 25992639
- [Derived] Van Dyke RB, Ngo-Giang-Huong N, Shapiro DE, Frenkel L, Britto P, Roongpisuthipong A, Beck IA, Yuthavisuthi P, Prommas S, Puthanakit T, Achalapong J, Chotivanich N, Rasri W, Cressey TR, Maupin R, Mirochnick M, Jourdain G; IMPAACT P1032 Protocol Team. A comparison of 3 regimens to prevent nevirapine resistance mutations in HIV-infected pregnant women receiving a single intrapartum dose of nevirapine. Clin Infect Dis. 2012 Jan 15;54(2):285-93. doi: 10.1093/cid/cir798. Epub 2011 Dec 5. PMID 22144539
- See also: Program for HIV Prevention and Treatment (PHPT), Thailand — http://www.phpt.org